CLINICAL TRIAL: NCT03165461
Title: Evaluation of the Use of Tracheal Intubation Through a Laryngeal Tube to Intubate Anesthetized Patients
Acronym: IKING
Status: Completed | Type: Observational
Sponsor: Formacion Internacional para la Docencia e Investigación de la Vía Aérea (Other)
Responsible Party: Principal Investigator, pedro charco mora, Director, Formacion Internacional para la Docencia e Investigación de la Vía Aérea
Other Study IDs: HCV2017LT
Record Dates: First submitted 2017-05-21; First posted 2017-05-24 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Airway Obstruction; Difficult Intubation
Keywords: intubation to supraglottic devices; intubating laryngeal tube
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Failed intubation is currently one of the most important factors leading to morbidity and mortality in anesthesia.

The development of supraglottic airway devices (SGDs), such as the intubating laryngeal tube, has revolutionized airway management, as these devices allow adequate ventilation and oxygenation in situations where ventilation and/or intubation via conventional means pose a challenge. Several publications describe the usefulness of such devices for salvaging ventilation in patients that cannot be intubated with direct laryngoscopy or who cannot be ventilated with a facemask. In these salvage situations, SGDs are highly effective in achieving adequate patient oxygenation.

Achieving effective oxygenation with an SGD and completely isolating the airway by intubation at the same time. This is now possible thanks to the so called supraglottic intubation devices (SGIDs). For that reason, we believe it is necessary to conduct a study that allows evaluation of the performance of this device in the context of daily clinical practice.

Its design characteristics, its capacity to be used in intubation applications, its soft and atraumatic materials as well as its disposability augur this product a significant expansion in the next few years. Nonetheless, no data are available on the success of intubation when the intubating laryngeal tube suction device (ILTSD) is used. The idea behind this study is to assess the possibilities to use the ITLSD device to intubate patients in regular anesthetic practice.

DETAILED DESCRIPTION:
The development of supraglottic airway devices (SGDs), such as the intubating laryngeal tube, has revolutionized airway management, as these devices allow adequate ventilation and oxygenation in situations where ventilation and/or intubation via conventional means pose a challenge. It would seem ideal to be able to unify both techniques in one single device; in other words, achieving effective oxygenation with an SGD and completely isolating the airway by intubation at the same time. This is now possible thanks to the so-called supraglottic intubation devices (SGIDs). For that reason, we believe it is necessary to conduct a study that allows evaluation of the performance of this device in the context of daily clinical practice.

LOCATION: The study will be conducted at operating rooms serving inpatients at the Valencia Clinical University Hospital. Investigators will be anesthesiologists with long experience in fibroscopy and in the management of supraglottic devices used for intubation.

METHODOLOGY: Prospective observational study aimed at evaluating the success of intubation through an I-LTSD device in regular clinical practice.

Research population: The study population will be made up of adult patients undergoing elective surgery who require general anesthesia and endotracheal intubation. Patients will be included in a consecutive manner provided that selection criteria are met. All patients will be required to sign an informed consent form.

Study variables: Information on the following variables will be gathered:

* Demographic variables: age, gender, weight, height
* Clinical variables: American Society Anaesthesiology status
* Concomitant conditions: presence of cardiovascular or respiratory conditions, liver or renal failure, history of gastroesophagic reflux.
* Type of surgery to be performed
* Difficult airway parameters:

  * Mallampati score
  * Thyromental distance
  * Degree of cervical mobility
  * Interdental distance (in mm)
* Anesthetic agents used, including dose administered: propofol, fentanyl, others
* Number of attempted laryngeal mask insertions
* Repositioning maneuvers
* Insertion time (in seconds)
* Change for a different number
* Expired tidal volume > 6-7 ml.kg-1,
* Expired CO2 < 45 mm Hg
* Seal pressure
* Fiberoptic visualization
* Ease of passage of nasogastric tube
* Number and duration of intubation attempts through laryngeal mask
* Presence of blood on removal of the device
* Soreness of throat, painful swallowing /intensity (mild-moderate-severe)
* Total anesthesia time
* Baseline hemodynamic parameters (SpO2, E-T-CO2) and BIS value at pre-insertion (following induction of anesthesia), at 3 minutes after insertion of I-LTSD device, pre-intubation and immediately following tube removal.

PATIENT RECRUITMENT Once it has been ascertained that inclusion criteria are met, patients will be informed about the study and they will be invited to participate. If they agree, they will be asked to sign an informed consent form either in the pre-anesthesia unit or in the ward. This must be done well before the patient is taken to the operating room.

OPERATION ROOM PROCEDURE (OR) Once the patient is in the OR standard monitoring is performed (3-lead ECG, non invasive blood pressure measurements every 5 minutes and peripheral O2 saturation). In addition, anesthetic depth will also be monitored using a bispectral index (BIS) monitor (BIS-VISTA™ Monitoring System, Aspect Medical System Inc. USA). Pre-oxygenation with 100% oxygen will be performed through a facemask with the patient breathing normally (normal tidal volume).

Subsequently the anesthesiologist in charge will carry out induction of anesthesia following the standard procedure, using neuromuscular blocking agents at standard doses (preferably rocuronium at a dose of 0.6 mg/kg of ideal weight). A record will be kept of the dosage used for each of the drugs administered during anesthesia induction. Once the patient has lost consciousness, manual ventilation will be applied through a facemask until the device is inserted.

According to airway management clinical guidelines,, anesthetic depth is considered adequate for insertion of a supraglottic device when the following conditions are met: absence of palpebral reflex, absence of response to jaw subluxation and BIS value below 40. If on insertion of the I-LTSD device the patient reacts with avoidance movements, the dose of propofol (or of the hypnotic agent the anesthetist in change has decided to use) should be augmented in 50 mg-bolus increments until the anesthetic status of the patient is appropriate for insertion of the device. A record will be kept of the total number of additional boluses required (if any).

The anesthesiologist will then insert the I-LTSD device in accordance with the manufacturer's instructions to ensure optimal placement:

* The size of the device is selected depending on the patient's ideal weight. Size 4-5 is recommended for adult patients (both males and females). A smaller size should be used in individuals whose weight or height is lower than the ideal value. .
* The anteroposterior and lateral surfaces of the I-LTSD device should be previously lubricated. Integrity of the device is checked by using the fingers to compress its distal portion (the area over the cuff). The device can be inserted with the head and neck placed in different positions, although the sniffing position is the most appropriate one.
* The device must be grasped with the dominant hand, with the thumb, index and middle fingers holding the base of the ventilation channel. Pressure is exerted posteriorly and caudally on the tube. The tube is inserted into the mouth passing the hard palate first and the soft palate later until it reaches its final position on the upper esophagic sphincter. Proper positioning of the device is indicated by resistance to its further advancement. Once the device is in place, soft manual ventilation must be performed to confirm it is in the proper position.
* Proper functioning of the I-LTSD device is confirmed by the absence of leakages, an initial tidal volume of 6-7 ml.kg-1, correct ventilatory chest movements and a normal expired CO2 curve. Should ventilation be ineffective, the anesthesiologist must reposition the device with maneuvers of the head, neck and jaw.

Once the I-LTSD device has been inserted:

* Airway quality is classified into: free, partially obstructed and fully obstructed. The existence of partial leaks will also be investigated. A maximum of three attempts will be allowed and, if necessary, recourse will be made to a different device or to standard intubation.
* The anatomical position of the I-LTSD device will be evaluated by fiberoptic visualization through the pneumatic cannel. Grade 1 corresponds to situations where the anterior epiglottis blocks visualization of the glottis or where laryngeal structures are absent. Grade 2 refers to cases where the anterior epiglottis and the vocal cords are visible. Grade 3 includes cases where the posterior epiglottis and the vocal cords can be seen. In grade 4 cases, full visualization of the vocal cords is possible. This assessment will be conducted by a different anesthesiologist from the one performing the intubation protocol.
* Seal pressure will be calculating in accordance with the methodology described above: the expiratory valve of the circle system must be closed at a constant fresh gas flow of 3 L/min, adjusting the pressure limiting valve to 40 cm H2O. Pressure in the circuit rises until equilibrium is reached and a leak is induced. That is the so-called seal pressure. Seal pressure will be determined 3-5 minutes after insertion, when it is functioning in a stable way. Audible leaks in the mouth, or reaching equilibrium, will determine the degree of seal pressure of the system.
* A record will be made of ease of passage of a 16 french nasogastric tube through the gastric channel (which will be previously lubricated and inserted only when the laryngeal tube is already in its final position).
* Once the laryngeal tube is in the ideal position, intubation can begin. An endotracheal tube (ETT) of the size recommended by the manufacturer will be used (a nr 7.5 ETT for a 4-5 I-LTSD device; a 7 ETT for a 2.5-3 I-LTSD device). If blind insertion of the ETT fails after two attempts and after correction maneuvers indicated by the anesthesiologist (removal a few centimeters of the laryngeal tube, rotating the ETT, anterior cervical movements,...), then intubation will be performed with a flexible fibroscope/endoscope and the study will be finalized.

Use of the fibroscope to facilitate endotracheal intubation is based on previous experience with these kinds of devices.

Training of the investigators in the procedures of the study:

The study will be carried out by physicians specializing in the fields of anesthesia and resuscitation who are in the habit of applying general anesthesia to patients undergoing surgery, and who routinely perform airway control by means of endotracheal intubation. They will also have used supraglottic devices for intubation in over 80 cases.

ESTIMATION SAMPLE SIZE& DATA ANALYSIS: According to published data, the success rate for other supraglottic devices ranges between 84 and 90% at the first attempt and between 95-100% overall. Considering that the upper limit of the 95% confidence interval acceptable for supraglottic devices should be lower than 2.5%, the required size of our sample should be of 30 patients. To compensate for potential losses to follow up, the total number of patients to be included will be 34.

The descriptive analysis of the data collected will be made by drawing up frequency tables for the nominal variables, and calculating measures of central tendency and dispersion for continuous variables. 95% confidence intervals will be estimated (95% CI) for the latter. For the clinical variables, Student's T test will be used for data related with quantitative variables if parameters show a normal distribution. If the distribution of parameters is abnormal the Mann-Whitney U test will be performed.

DURATION: The data recording period will be 5 months. Patients will be recruited consecutively provided that they comply with the inclusion criteria, they do not meet the exclusion criteria described above and they agree to participate in the study and sign the required informed consent form.

ETHICAL: The study will be conducted in accordance with the ethical requirements laid down in the Helsinki Declaration, revised in Edinburgh, Scotland in October 2000, in terms of human experimentation, as well as in accordance to Spanish Royal Decree 223 of 1 May 2004.

CONFIDENTIALITY: The study will be carried out within the framework of the Spanish Data Protection Law (Act 15 of 13 December 1999).

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II & III.
* Age over 18.
* Outpatient and inpatient surgery requiring endotracheal intubation. Signature of an informed consent form.

Exclusion Criteria:

* Patients who, on initial airway examination, exhibit any of the following conditions associated with a difficult airway: cervical spine pathology, mouth opening restriction of less than 3 cm. (combination of Mallampati class III-IV, thyromental distance < 6 cm and reduced mouth opening).
* A history of severe gastroesophagic reflux and/or a history of recent respiratory infection.
* Refusal of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of adult patients undergoing elective surgery who require general anesthesia and endotracheal intubation. Patients will be included in a consecutive manner provided that selection criteria are met, then patients will be informed about the study and they will be invited to participate. If they agree, they will be asked to sign an informed consent form either in the pre-anesthesia unit or in the ward. This must be done well before the patient is taken to the operating room.
  All patients will be required to sign an informed consent form.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluate success of fiberoptic guide endotraqueal intubation through an I-LTSD device in patients to general anesthesia without difficult intubation. | one day
  The study will determinate the success of visual fiberoptic intubation at a first and a second attempt and guided fiberoptic intubation at a third and last attempt. Should the third attempt fail, intubation will be performed through direct or indirect laryngoscopy.
  The initial success rate will be calculated and the number of attempts needed for successful intubation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: pedro Charco-Mora, MD, PhD, Study Chair — Formacion Internacional para la Docencia e Investigación de la Vía Aérea
Locations (1):
- Pedro Charco Mora, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergold MN, Kahle S, Schultzik T, Bucheler M, Byhahn C. [Intubating laryngeal tube suction disposable: Initial clinical experiences with a novel device for endotracheal intubation]. Anaesthesist. 2016 Jan;65(1):30-35. doi: 10.1007/s00101-015-0100-0. Epub 2015 Oct 19. German. PMID 26481391
- [Result] Landsdalen HE, Berge M, Kristensen F, Guttormsen AB, Softeland E. Continuous ventilation during intubation through a supraglottic airway device guided by fiberoptic bronchoscopy: a observational assessment. Acta Anaesthesiol Scand. 2017 Jan;61(1):23-30. doi: 10.1111/aas.12824. Epub 2016 Nov 3. PMID 27808401
- [Result] Michalek P, Donaldson W, McAleavey F, Abraham A, Mathers RJ, Telford C. The i-gel Supraglottic Airway as a Conduit for Fibreoptic Tracheal Intubation - A Randomized Comparison with the Single-use Intubating Laryngeal Mask Airway and CTrach Laryngeal Mask in Patients with Predicted Difficult Laryngoscopy. Prague Med Rep. 2016;117(4):164-175. doi: 10.14712/23362936.2016.17. PMID 27930894
- [Result] Metterlein T, Dintenfelder A, Plank C, Graf B, Roth G. A comparison of various supraglottic airway devices for fiberoptical guided tracheal intubation. Braz J Anesthesiol. 2017 Mar-Apr;67(2):166-171. doi: 10.1016/j.bjane.2015.09.007. Epub 2016 May 26. PMID 28236864